CLINICAL TRIAL: NCT03697174
Title: Acute Health Effects of Ozone Exposure in Healthy Young Adults: a Randomized Controlled Study
Brief Title: Acute Health Effects of Ozone Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haidong Kan, Professor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: FDUEH-5
Record Dates: First submitted 2018-09-30; First posted 2018-10-05 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Function

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure group (Experimental): Subjects in exposure group will be exposed to 200 ppb ozone for 2 hours in a chamber.
  Interventions: Other: 200 ppb ozone group
- Control group (Sham Comparator): Subjects in control group will be exposed to 0 ppb ozone (clean air) for 2 hours in a chamber.
  Interventions: Other: 0 ppb ozone group

INTERVENTIONS:
Other: 200 ppb ozone group — The exposure group will be exposed to 200 ppb ozone in a chamber for 2 hours while alternating 20-min rest and 10-min exercise periods. The exercise workload will be adjusted to achieve the targeted ventilation of 25 ~ 27 L/min(approximately equal to 15 ~ 18L/min/m2 body surface area). The temperature and relative humidity in the chamber will be maintained at 22±1℃ and 55%±5%, respectively.
  Arms: Exposure group
Other: 0 ppb ozone group — The control group will be exposed to 0 ppb ozone in a chamber for 2 hours while alternating 20-min rest and 10-min exercise periods. The exercise workload will be adjusted to achieve the targeted ventilation of 25 ~ 27 L/min(approximately equal to 15 ~ 18L/min/m2 body surface area). The temperature and relative humidity in the chamber will be maintained at 22±1℃ and 55%±5%, respectively.
  Arms: Control group

SUMMARY:
This is a randomized controlled human exposure crossover study. Investigators aim to investigate the acute health effects of ozone exposure in healthy young adults.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled human exposure crossover study among 32 healthy young adults in Shanghai, China. Each subject will be exposed twice: once to clean air and once to 200 ppb ozone in a chamber for 2 hours. During the 2-hour exposure, each subject will be requested to alternate 20 minutes of rest and 10 minutes of exercise on a treadmill. The exercise workload will be adjusted to achieve the targeted ventilation of 25 ~ 27 L/min(approximately equal to 15 ~ 18L/min/m2 body surface area). Ozone will be generated by a silent electric discharge method (HTU-500, AZCO Industries Ltd., Canada) and introduced into the chamber. The temperature and relative humidity in the chamber will be maintained at 22±1℃ and 55%±5%, respectively. Health examinations will be conducted immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning. Health examinations include symptom questionnaire, skin tests, spirometry, and Holter monitoring. We plan to collect blood, buccal, urine, nasal secretion, saliva, exhaled breath condensate, sebum, and D-squame samples.

ELIGIBILITY:
Inclusion Criteria:

* Living in Shanghai during study period;
* Ability to complete the exercise to achieve the ventilation of 15 to 18 L/min/m2 body surface area;
* Body mass index >18.5 and ≤30.0 (30 is the lower limit for class 2 obesity for Chinese).

Exclusion Criteria:

* Smoking and alcohol abuse;
* Current drug and dietary supplements intake;
* Subjects with allergic diseases, such as allergic rhinitis, allergic asthma, and atopy;
* Subjects with cardiovascular diseases, such as congenital heart disease, pulmonary heart disease, and hypertension;
* Subjects with respiratory diseases, such as asthma, chronic bronchitis, and chronic obstructive pulmonary disease;
* Subjects with chronic diseases, such as diabetes, chronic hepatitis, and kidney disease;
* Subjects who have a history of major surgery;
* Abnormal spirometry (FEV1 and FVC ≤ 75% of predicted and FEV1/FVC ≤ 0.65);
* Abnormal baseline 12-lead resting electrocardiogram;
* Abnormal blood index, such as cell counting, blood lipids, and glutamic-pyruvic transaminase (GPT).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2018-12-09 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
Changes of FEV1 | FEV1 will be examined immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning
  Changes of forced expiratory volume in 1 second
Changes of FVC | FVC will be examined immediately prior to exposure, immediately after exposure, 2 hours after exposure and again the next morning
  Changes of forced vital capacity

SECONDARY OUTCOMES:
HRV | Holter monitoring will be performed continuously for 24 hours.
  Heart rate variability

OTHER OUTCOMES:
Difference in CRF concentrations between the two exposures | 2 hours after the completion of exposure.
  Difference in the serum concentrations of corticotrophin releasing factor between ozone exposure and filtered air exposure
Difference in ACTH concentrations between the two exposures | 2 hours after the completion of exposure.
  Difference in the serum concentrations of adrenocorticotropic hormone between ozone exposure and filtered air exposure
Difference in cortisol concentrations between the two exposures | 2 hours after the completion of exposure
  Difference in the serum concentrations of cortisol between ozone exposure and filtered air exposure
Difference in adrenaline concentrations between the two exposures | 2 hours after the completion of exposure.
  Difference in the serum concentrations of adrenaline between ozone exposure and filtered air exposure
Difference in noradrenaline concentrations between the two exposures | 2 hours after the completion of exposure.
  Difference in the serum concentrations of noradrenaline between ozone exposure and filtered air exposure
Change in the amount of skin moisture | Immediately before exposure, 0.5 hours after the completion of exposure, and next morning.
  Change in the amount of skin moisture, which was measure by a moisture meter. The number on the meter indicates how hydrated (or dehydrated) your skin is.
Change in L-values | Immediately before exposure, 0.5 hours after the completion of exposure, and next morning.
  Change in skin color indicated by L-values, which was measured by a skin colorimeter.
Change in a-values | Immediately before exposure, 0.5 hours after the completion of exposure, and next morning.
  Change in skin color indicated by a-values, which was measured by a skin colorimeter.
Change in b-values | Immediately before exposure, 0.5 hours after the completion of exposure, and next morning.
  Change in skin color indicated by b-values, which was measured by a skin colorimeter.
Difference in alpha diversity of microbiota between the two exposures | Immediately after the completion of exposure
  Difference in alpha diversity of microbiota in nasal secretions between ozone exposure and filtered air exposure
Change in CC16 concentrations | Immediately before exposure, 2 hours after the completion of exposure, and next morning
  Change in the serum concentrations of club cell protein
Differences in metabolite levels detected in serum metabolomics between the two exposures | 2 hours after the completion of exposure
  Mass spectrometry-based serum metabolomics is non-targeted.The study is to find the differential metabolites in serum between ozone exposure and filtered air exposure.
Differences in metabolite levels detected in airway metabolomics between the two exposures | 2 hours after the completion of exposure
  Mass spectrometry-based metabolomics in exhaled breath condensate is non-targeted.The study is to find the differential metabolites in airway between ozone exposure and filtered air exposure.
Differences in metabolite levels detected in urine metabolomics between the two exposures | Immediately after the completion of exposure
  Mass spectrometry-based urine metabolomics is non-targeted.The study is to find the differential metabolites in urine between ozone exposure and filtered air exposure.
Differences in RNA expression levels detected in transcriptomics between the two exposures | 2 hours after the completion of exposure
  Illumina-based transcriptomics is non-targeted. The study is to find the differentially expressed RNA between ozone exposure and filtered air exposure.
Differences in protein levels detected in serum proteomics between the two exposures | 2 hours after the completion of exposure
  Mass spectrometry-based proteomics in serum is non-targeted. The study is to find the differentially expressed proteins in serum between ozone exposure and filtered air exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Haidong Kan, Ph.D, Principal Investigator — Department of Environmental Health, School of Public Health, Fudan University
Locations (1):
- Department of Environmental Health, School of Public Health, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Niu Y, Chen R, Wang C, Wang W, Jiang J, Wu W, Cai J, Zhao Z, Xu X, Kan H. Ozone exposure leads to changes in airway permeability, microbiota and metabolome: a randomised, double-blind, crossover trial. Eur Respir J. 2020 Sep 3;56(3):2000165. doi: 10.1183/13993003.00165-2020. Print 2020 Sep. No abstract available. PMID 32299865